CLINICAL TRIAL: NCT00405457
Title: Efficacy and Safety of a New Multi-dose Lubricant Eye Drop Concomitant With Restasis® (Cyclosporine A) for the Treatment of Dry Eye Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: David Hardten, MD, Minnesota Eye Consultants
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5261
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

ARMS (1):
- A (Other)
  Interventions: Drug: Restasis, Optive Tears

INTERVENTIONS:
Drug: Restasis, Optive Tears — Restasis and Optive Tears use twice daily more frequently if needed

SUMMARY:
To evaluate the efficacy, safety and tolerability of a combination of Optive® Artificial Tears with Restasis®.The primary hypothesis is that the Ocular Surface Disease Index (OSDI) score and symptoms will be the same or lower than baseline after treatment in these patients. The patients will tolerate the combination of Restasis® and Optive® with a low incidence of clinical adverse events.

ELIGIBILITY:
Inclusion Criteria:

* · Males or females > 18 years old

  * Patients currently taking Restasis® for at least 3 months in duration and using artificial tears as needed for dry eye.
  * Likely to complete all study visits and able to provide informed consent

Exclusion Criteria:

* · Patients using Restasis® for less than 3 months.

  * Known contraindications to any study medication or ingredients
  * Female of child bearing potential not using reliable methods of birth control, or pregnant or lactating females.
  * Other active uncontrolled ocular diseases or uncontrolled systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
efficacy | 1 yr 3 months

SECONDARY OUTCOMES:
dry eye symptoms | 1 yr 3 months

CONTACTS AND LOCATIONS:
Overall Officials: David Hardten, MD, Principal Investigator — Minnesota Eye Consultants
Locations (1):
- Minnesota Eye Consultants, Minneapolis, Minnesota, United States